CLINICAL TRIAL: NCT06592898
Title: Different Squatting Modes in the Rehabilitation of Patellofemoral Pain Syndrome:A Prospective Randomized Controlled Trial
Brief Title: Different Squatting Modes in the Rehabilitation of Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2023013
Record Dates: First submitted 2024-07-25; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; static squat; rehabilitation
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group: straight leg raise (Active Comparator): The patient was supine position, one knee angle was 90°, the foot was flatted on the ground. The ankle was flexed to contract the quadriceps on the other side. Then straighten the knee joint and the hip was 30° and lift the thigh, the heel was about 20cm away from the ground, and put down the lower limb after 2 seconds. Ten times are in a group, each practice has 5 groups, rest between the groups is 1 minute. Practice 5 times a week, practice on both sides, take uniform respiration without holding breath.
  Interventions: Behavioral: straight leg raise
- Experimental group A: wall squat (Experimental): The subjects' upper body was upright, the distance between feet was same as width of shoulder, and hands were placed on each side of the body or above the thighs. Tiptoes were towards the front, and perpendicular to the wall. The distance between the wall and heel was about a foot long, and the back was close to the wall, squatted slowly.
  Interventions: Behavioral: wall squat
- Experimental group B: direct squat (Experimental): The subjects stood on the flat ground, the upper body was upright, the distance between feet was same as width of shoulder, and tiptoes were towards the front. The trunk was adjusted forward according to the Angle of static squat. The specific method is to adjust the trunk position to the line of the shoulder joint and knee joint perpendicular to the ground. Knee joint can bend at a large angle.The center of gravity was between the feet, put hands in front of body.The angle was set at 30° for the first two weeks, increased to 45° after two weeks, and set at 60° for the last two weeks.
  Interventions: Behavioral: direct squat
- Experimental group C: wall squat assisted by elastic bands (Experimental): Based on wall squat, subjects put elastic band of 20 pounds between the thighs, open thighs and feet at a low speed, so that the elastic bands were slightly deformed and sence of resistance was obvious on the outside of the thighs.The angle was set at 30° for the first two weeks, increased to 45° after two weeks, and set at 60° for the last two weeks.
  Interventions: Behavioral: wall squat assisted by elastic bands

INTERVENTIONS:
Behavioral: straight leg raise — The patient was supine position, one knee angle was 90°, the foot was flatted on the ground. The ankle was flexed to contract the quadriceps on the other side. Then straighten the knee joint and the hip was 30° and lift the thigh, the heel was about 20cm away from the ground, and put down the lower limb after 2 seconds. Ten times are in a group, each practice has 5 groups, rest between the groups is 1 minute. Practice 5 times a week, practice on both sides, take uniform respiration without holding breath.
  Arms: Control group: straight leg raise
Behavioral: wall squat — The subjects' upper body was upright, the distance between feet was same as width of shoulder, and hands were placed on each side of the body or above the thighs. Tiptoes were towards the front, and perpendicular to the wall. The distance between the wall and heel was about a foot long, and the back was close to the wall, squatted slowly.
  Arms: Experimental group A: wall squat
Behavioral: direct squat — The subjects stood on the flat ground, the upper body was upright, the distance between feet was same as width of shoulder, and tiptoes were towards the front. The trunk was adjusted forward according to the Angle of static squat. The specific method is to adjust the trunk position to the line of the shoulder joint and knee joint perpendicular to the ground. Knee joint can bend at a large angle. The center of gravity was between the feet, put hands in front of body.The angle was set at 30° for the first two weeks, increased to 45° after two weeks, and set at 60° for the last two weeks.
  Arms: Experimental group B: direct squat
Behavioral: wall squat assisted by elastic bands — Based on wall squat, subjects put elastic band of 20 pounds between the thighs, open thighs and feet at a low speed, so that the elastic bands were slightly deformed and sence of resistance was obvious on the outside of the thighs.The angle was set at 30° for the first two weeks, increased to 45° after two weeks, and set at 60° for the last two weeks.
  Arms: Experimental group C: wall squat assisted by elastic bands

SUMMARY:
This study take 84 patients with Patellofemoral Pain Syndrome in Peking University Third Hospital during January to September in 2023 as subjects, aiming to explore the efficacy and intervention effects of three different static squat modes including straight leg raise, wall squat, direct squat and wall squat assisted by elastic bands for patients with PFPS, in order to providing theoretical basis and effective guidance for future home rehabilitation of patients with PFPS combined with mobile health.

DETAILED DESCRIPTION:
Background：Static squat has been widely used in the treatments of patellofemoral pain syndrome (PFPS), but no study has assessed which static squat modes is more effective .This study aimed to compare the effects of three different static squat modes on patients with patellofemoral pain syndrome .

Methods：Investigators included 84 patients with patellofemoral pain syndrome, a 6-week training period using a mobile phone app with angle recognition function, patients were devided into 4 groups based on different static squat modes. Kujala score, Lysholm score, VAS-W score, VAS-U score,thigh circumference, peak torque of knee extension, and peak torque of knee flexion on the affected side were used to assess efficacy.Two-way ANOVA was conducted to determine the differences within and between groups.Paired-samples t-test was used for intergroup comparisons, and one-way ANOVA was applied for intergroup comparisons. Chi-square tests were performed on categorical data.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of PFPS.

  * Age between 20 and 45 years (to reduce the risk of suffer from patellofemoral joint bone joint)

    * Have no other treatments before the experiment.

      * Sign the informed consent form.

Exclusion Criteria:

* Patients with a history of knee surgery.

  * With other lower limb injuries such as meniscus tear, bursitis, ligament injury, patellar tendon injury, joint degeneration, etc.

    * With a history of dislocation and subluxation of patellofemoral joint.

      * With cardiovascular vessels, lung, kidney and other important organs.

        * Not available to use mobile phone APP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of three different static squat modes for home rehabilitation of patients with patellofemoral pain syndrome. | 6 weeks
  Investigators assessed the efficacy of wall squat, direct squat and wall squat assisted by elastic bands by measure Kujala score, Lysholm score, VAS-W score, VAS-U score, thigh circumference score, results of peak knee torque in isokinetic muscle strength test and peak knee moment results for isokinetic muscle strength test by using USA Biodex isokinetic muscle strength tester at 3rd week and 6th week. Before statistics, the measurement data are tested for normality and homogeneity of variance. The data meet the conditions of normal distribution and homogeneity of variance, and the statistical results are expressed in the form of mean ± standard deviation (x ± s).Count data were analyzed by the chi-square test. P <0.05 represents a statistically significant difference.
  Higher values for all scores proved better intervention treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No